CLINICAL TRIAL: NCT02001480
Title: Surrogate Markers for Sudden Cardiac Death in Patients With Diabetes Mellitus and End Stage Renal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-039
Record Dates: First submitted 2013-10-23; First posted 2013-12-05 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus Type 2; End Stage Renal Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Failure, Chronic | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Echocardiography (Other): 12 lead holter for 7 days
  CGM = continuous Glucose Monitoring
  Interventions: Device: 12 lead Holter; Device: CGM Continuous Glucose Monitoring

INTERVENTIONS:
Device: 12 lead Holter — 12 lead Holter measurements will be performed for 7 days
Device: CGM Continuous Glucose Monitoring — CGM will be performed continously for 7 days

SUMMARY:
Aim: Patients with type 2 diabetes mellitus (T2DM) and hemodialysis due to diabetic nephropathy exhibit a high risk for sudden cardiac death (SCD). Preliminary data suggest that beta-blocker treatment may reduce arrhythmias and mortality in this high-risk population. However, no results from large-scale clinical outcome trials with beta-blockers exist in this patient group and a broad, scientifically unapproved use of beta-blocker treatment may not be justified due to potential harmful side-effects such as AV-block or hypotension. In addition, we are lacking identified ECG surrogate parameters for SCD in this high-risk population and on the occurrence of arrhythmias in temporary relationship to hemodialysis sessions.

Therefore, the present study will identify surrogate parameters of SCD in hemodialysis patients with T2DM and in an interventional trial investigate the suppressive effect of beta-blockers on these identified ECG markers.

ELIGIBILITY:
Inclusion Criteria:

* patients with diabetes mellitus type 2
* chronic hemodialysis at least since 3 months
* aged above 18 years
* written informed consent
* legally competent

Exclusion Criteria:

* intake of bets-blockker within the last four weeks
* pregnancy and breast feeding
* abuse of drugs and alcohol
* missing compliance
* life expectancy < 6 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
ECG surrogate markers compared to cardiac events | Analysis will be performed after last patient is out
  Recruiting Period: October 2013 - April 2014 (6 months)/ Last patient out: April 2014/ Data cleaning, processing, analysis, study report: May 2014 - October 2014 (6 months)

SECONDARY OUTCOMES:
Continuous glucose monitoring is performed to identify episodes of hypoglycaemia | Analysis will be done after last patient is out
  Recruiting/active Period: October 2013 - April 2014 (6 months)/ Last patient out: April 2014/ Data cleaning, processing, analysis, study report: May 2014 - October 2014 (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Marx, Univ.-Prof., Principal Investigator — Department of Internal Medicine University Hospital Aachen
Locations (3):
- Germany (3):
  - regioMed-Kliniken GmbH, Coburg, Bavaria
  - University Hospital Würzburg, Würzburg, Bavaria
  - Department of Internal Medicine I University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia